CLINICAL TRIAL: NCT01273558
Title: An Open-Label Study to Compare Two Methods for Determining the Renal Threshold for Glucose in Subjects With Type 2 Diabetes Mellitus
Brief Title: A Study of Two Methods for Determining the Renal Threshold for Glucose in Patients With Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Responsible Party: Sponsor
Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR017719; 28431754DIA1025 (Other: Johnson & Johnson Pharmaceutical Research & Development, L.L.C.)
Record Dates: First submitted 2010-12-10; First posted 2011-01-10 (Estimated); Last update posted 2013-04-22 (Estimated); Status verified 2013-04

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Canagliflozin; Renal threshold for glucose; Pharmacodynamics
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Canagliflozin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Part 1: no Intervention (No Intervention): In Part 1 of the study, patients will not receive any study drug.
- Part 2: canagliflozin (Experimental): In Part 2 of the study, patients will receive canagliflozin once daily on Days 1 through 8.
  Interventions: Drug: Canagliflozin

INTERVENTIONS:
Drug: Canagliflozin — One 100 mg capsule taken orally (by mouth) on Days Days 1-8
  Arms: Part 2: canagliflozin

SUMMARY:
The purpose of this study is to compare the results from two methods used to determine the renal threshold for glucose excretion (defined as the lowest plasma glucose concentration at which appreciable amounts of glucose appear in the urine) in untreated patients with type 2 diabetes mellitus and in patients with type 2 diabetes mellitus who are treated with 100 mg once-daily canigliflozin for 8 days.

DETAILED DESCRIPTION:
This is an open-label (patients will know if they are receiving treatment and the identity of the treatment) study that will compare renal threshold of glucose (RTG) values obtained by 2 different methods: an established method (ie, the stepwise hyperglycemic clamp method) and a new method (the mixed meal tolerance test [MMTT] method). The RTG is defined as the lowest plasma glucose concentration at which appreciable amounts of glucose appear in the urine. Each method for determining the RTG value will be performed in untreated patients with type 2 diabetes mellitus (T2DM) and in patients with T2DM who are treated with canagliflozin 100 mg once daily for 8 days. Canagliflozin (a Sodium-Glucose Cotransporter 2 inhibitor) is currently under development to lower blood sugar levels in patients with T2DM. Patients will not take study drug (canagliflozin 100 mg overencapsulated tablets) in Part 1 of the study. In Part 2 of the study, patients will take study drug once daily on Study Days 1 through 8.

ELIGIBILITY:
Inclusion Criteria:

* Patients with T2DM who are not receiving treatment with any anti-hyperglycemic agents (AHAs) for at least 12 weeks, or who are receiving treatment with a stable dose and regimen of metformin monotherapy for at least 12 weeks and have a hemoglobin A1c (HbA1c) in the range of >=7% to <=10%

Exclusion Criteria:

* History of Type 1, "brittle" diabetes or secondary forms of diabetes
* History of 1 or more severe hypoglycemic episodes
* History of diabetic complications considered to be clinically significant by the Investigator
* History of or current illness considered to be clinically significant by the investigator

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2011-01; Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
RTG values using the MMTT and the stepwise hyperglycemic clamp methods | On Days 1 and 2 (Part 1)
RTG values using the MMTT and the stepwise hyperglycemic clamp methods | On Days 7 and 8 (Part 2)

SECONDARY OUTCOMES:
Plasma glucose (PG) concentration during the MMT and the hyperglycemic clamp procedure | On Days 1 and 2 (Part 1)
Plasma glucose (PG) concentration during the MMT and the hyperglycemic clamp procedure | On Days 7 and 8 (Part 2)
Rate of Urinary glucose excretion (UGE) during the MMTT and the hyperglycemic clamp procedure | On Days 1 and 2 (Part 1)
Rate of Urinary glucose excretion (UGE) during the MMTT and the hyperglycemic clamp procedure | On Days 7 and 8 (Part 2)

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.
Locations (1):
- Neuss, Germany

REFERENCES:
- [Derived] Polidori D, Sha S, Ghosh A, Plum-Morschel L, Heise T, Rothenberg P. Validation of a novel method for determining the renal threshold for glucose excretion in untreated and canagliflozin-treated subjects with type 2 diabetes mellitus. J Clin Endocrinol Metab. 2013 May;98(5):E867-71. doi: 10.1210/jc.2012-4205. Epub 2013 Apr 12. PMID 23585665
- See also: An Open-Label Study to Compare Two Methods for Determining the Renal Threshold for Glucose in Subjects With Type 2 Diabetes Mellitus — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=877&filename=CR017719_CSR.pdf